CLINICAL TRIAL: NCT02151903
Title: An Open-Label Extension Study of De-immunized DI-Leu16-IL2 Immunocytokine Administered in Patients With B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Open-Label Extension Study of De-immunized DI-Leu16-IL2 Immunocytokine Administered in Participants With B-cell NHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical benefit was noted before the scheduled completion of the trial and the extension study was terminated early.
Sponsor: Alopexx Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AO-101-EXT
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: NHL; Immunocytokine; Lymphoma; Non-Hodgkin; B-cell; IL (interleukin)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DI-Leu16-IL2 1.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 1.0 milligrams per square meter (mg/m^2) subcutaneously (SC) for 3 consecutive days every 3 weeks (21-day cycle). Participants will continue to receive therapy through the duration of the study as long as they will have clinical benefit and will not experience any untoward side effects.
  Interventions: Drug: DI-Leu16-IL2
- DI-Leu16-IL2 2.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 2.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle). Participants will continue to receive therapy through the duration of the study as long as they will have clinical benefit and will not experience any untoward side effects.
  Interventions: Drug: DI-Leu16-IL2

INTERVENTIONS:
Drug: DI-Leu16-IL2 — DI-Leu16-IL2 will be administered per dose and schedule specified in the arm.

SUMMARY:
This is an open-label extension study enrolling participants experiencing clinical benefit following 6 cycles of DI-Leu16-IL2 while enrolled in the Alopexx Oncology Dose-Escalation AO-101 study (NCT01874288). Participants will be permitted to continue to receive DI-Leu16-IL2 at the same dose, schedule, and route of administration they received during Study AO-101 (Main Study). Prior pre-treatment (for example, Rituximab) will continue as before.

ELIGIBILITY:
Inclusion Criteria:

1. Participants currently entered on Alopexx Oncology Study AO-101
2. Participants who received 6 cycles of DI-Leu16-IL2 on Study AO-101.
3. Documented clinical benefit following 6th cycle of DI-Leu16-IL2
4. Able to begin extension study within 8 weeks of receiving 6th cycle of DI-Leu16-IL2
5. Participants must have received prior Rituximab-containing therapy.
6. Participants in this extension study are to use adequate birth control measures (abstinence, oral contraceptives, barrier method with spermicide or surgical sterilization) during the study. Females of childbearing potential must have a negative serum pregnancy test on the days of dosing. A female of childbearing potential: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (that is, has had menses at any time in the preceding 24 consecutive months.
7. Provide written informed consent prior to any study procedures.

Exclusion Criteria:

1. Pregnant or lactating female
2. An immediate need for palliative radiotherapy or systemic corticosteroid therapy.
3. Actively infected with or chronic carriers of hepatitis B virus (HBV) as demonstrated by positive hepatitis B core antibody (HbcAb) or hepatitis B surface antigen (HbsAg). Participants who are sero-positive only, that is, surface antibody positive [HbsAb], are permitted.
4. Other significant active infection
5. Major surgery, chemotherapy, investigational agent, or radiation within 30 days of Day 1
6. Uncontrolled hypertension (diastolic ≥ 100 millimeters of mercury [mmHg]) or hypotension (systolic ≤ 90 mmHg)
7. History of prior therapy or a serious, uncontrolled medical disorder that in the Investigator's opinion would impair participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Vlock, MD, Study Director — Alopexx Oncology, LLC
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] Ko YJ, Bubley GJ, Weber R, Redfern C, Gold DP, Finke L, Kovar A, Dahl T, Gillies SD. Safety, pharmacokinetics, and biological pharmacodynamics of the immunocytokine EMD 273066 (huKS-IL2): results of a phase I trial in patients with prostate cancer. J Immunother. 2004 May-Jun;27(3):232-9. doi: 10.1097/00002371-200405000-00008. PMID 15076141
- [Background] King DM, Albertini MR, Schalch H, Hank JA, Gan J, Surfus J, Mahvi D, Schiller JH, Warner T, Kim K, Eickhoff J, Kendra K, Reisfeld R, Gillies SD, Sondel P. Phase I clinical trial of the immunocytokine EMD 273063 in melanoma patients. J Clin Oncol. 2004 Nov 15;22(22):4463-73. doi: 10.1200/JCO.2004.11.035. Epub 2004 Oct 13. PMID 15483010
- [Background] Maloney DG, Liles TM, Czerwinski DK, Waldichuk C, Rosenberg J, Grillo-Lopez A, Levy R. Phase I clinical trial using escalating single-dose infusion of chimeric anti-CD20 monoclonal antibody (IDEC-C2B8) in patients with recurrent B-cell lymphoma. Blood. 1994 Oct 15;84(8):2457-66. PMID 7522629
- See also: Sponsor website — http://www.alopexx.com
- See also: National Cancer Institute at the National Institute of Health — http://www.cancer.gov/cancertopics/types/non-hodgkin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who, in the opinion of the Investigator, exhibited a beneficial effect without a dose-limiting toxicity (DLT) in the dose-escalation Study AO-101 (NCT01874288) (Main Study) were allowed to continue treatment with DI-Leu16-IL2 in this open-label extension study.
Groups:
- DI-Leu16-IL2 1.0 mg/m^2: Participants received DI-Leu16-IL2 1.0 milligrams per square meter (mg/m^2) subcutaneously (SC) for 3 consecutive days every 3 weeks (21-day cycle). Participants continued to receive therapy through the duration of the study as long as they were having clinical benefit and not experiencing any untoward side effects.
- DI-Leu16-IL2 2.0 mg/m^2: Participants received DI-Leu16-IL2 2.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle). Participants continued to receive therapy through the duration of the study as long as they were having clinical benefit and not experiencing any untoward side effects.
Period: Overall Study
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Started | 3 | 2
Received at Least 1 Dose of Study Drug | 3 | 2
Completed | 0 | 1
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Progressive disease | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- DI-Leu16-IL2 1.0 mg/m^2: Participants received DI-Leu16-IL2 1.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle). Participants continued to receive therapy through the duration of the study as long as they were having clinical benefit and not experiencing any untoward side effects.
- Total: Total of all reporting groups
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Overall Response (BOR) Assessed Per International Workshop for Non-Hodgkin Lymphoma (NHL) Response Criteria
Description: BOR included complete response (CR), unconfirmed CR (CRu), partial response (PR), stable disease (SD), and progressive disease (PD). CR: 1)Disappearance of all detectable clinical and radiological evidence of disease; 2)lymph nodes (LN) regressed to normal size; 3)other organs (spleen, liver, kidneys) that were enlarged before therapy must have decreased in size; 4)clear bone marrow(BM) infiltrate. CRu: must meet CR criteria 1 and 3, as well as ≥1 of following: residual LN mass >1.5 centimeters (cm) in greatest transverse diameter; individual nodes that were previously confluent regressed by >75% in sum of product diameters (SPD); or indeterminate BM. PR: 6 largest dominant nodes or nodal masses decreased by ≤50% in SPD; no increase in size of other nodes; liver or spleen; splenic and hepatic nodules regressed ≥50% in SPD; and no new disease. SD: less than a PR but not PD. PD: 50% increase from nadir in SPD of any abnormal node for PR or nonresponders and appearance of any new lesion.
Time Frame: First dose of study drug until first appearance of CR, CRu, PR, SD, or PD (up to 20 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 3 | 2
Participants
  CR | 0 | 1
  CRu | 0 | 0
  PR | 0 | 0
  SD | 1 | 0
  PD | 1 | 1

2. Primary Outcome: Tumor Measurement: Percent Change From Baseline in Sum of Product of Diameters at the End of Study
Description: Sum of product diameters sums the product of the 2 tumor measurements on each lesion. If only 1 measurement was available, it was used as the longest length and the product of the lengths in the sum. Baseline value is the last non-missing measurement prior to receiving study drug injection in the Main Study AO-101.
Time Frame: Baseline, end of study (EOS) (up to approximately 32 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. None of the participants were considered evaluable in 'DI-Leu16-IL2 2.0 mg/m^2' arm for this outcome measure at the end of study, and therefore, data were not collected for that arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 2 | 0
percent change | -22.86066 (9.805965) |

3. Primary Outcome: Tumor Measurement: Percent Change From Baseline in Sum of Longest Diameters at the End of Study
Description: Sum of longest diameters is the sum of the longest measured length of each tumor lesion. Baseline value is the last non-missing measurement prior to receiving study drug injection in the Main Study AO-101. None of the participants were considered evaluable in 'DI-Leu16-IL2 2.0 mg/m^2' arm for this outcome measure at the end of study, and therefore, data were not collected for that arm
Time Frame: Baseline, EOS (up to approximately 32 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 2 | 0
percent change | -11.638 (1.5001) |

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs with onset at the time of or following the start of treatment with study drug, or AEs starting before the start of treatment but increasing in severity or relationship at the time of or following the start of treatment. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: First dose of study drug up to EOS (up to 20 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 3 | 2
Participants
  Any TEAEs | 3 | 1
  SAEs | 2 | 0

5. Secondary Outcome: Number of Participants With a TEAE That Was Considered Related to a Clinically Significant Hematology or Serum Chemistry Abnormality
Description: TEAEs were defined as AEs with onset at the time of or following the start of treatment with study drug, or AEs starting before the start of treatment but increasing in severity or relationship at the time of or following the start of treatment. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Clinically significant hematology and serum chemistry abnormalities were identified at the Investigator's discretion.
Time Frame: First dose of study drug up to EOS (up to 20 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 3 | 2
Participants | 3 | 0

6. Secondary Outcome: Number of Participants With a Clinically Significant Abnormal Physical Exam
Description: Clinically significant abnormal physical exams included extremities, head, ears, eyes, nose, throat, abdomen, respiratory system, lymphatic system, and integumentary system. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. Clinically significant abnormal physical exams were identified at the Investigator's discretion.
Time Frame: First dose of study drug up to EOS (up to 20 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
Number analyzed (Participants) | 3 | 2
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: First dose of study drug up to EOS (up to 20 months)
Description: Safety population included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DI-Leu16-IL2 1.0 mg/m^2 (N=3) | DI-Leu16-IL2 2.0 mg/m^2 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DI-Leu16-IL2 1.0 mg/m^2 (N=3) | DI-Leu16-IL2 2.0 mg/m^2 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 1
Injection site induration (General disorders) | 1 | 1
Injection site oedema (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Hematocrit decreased (Investigations) | 1 | 0
Protein total increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 1
Injection site swelling (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Injection site inflammation (General disorders) | 0 | 1
Injection site mass (General disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Clinical benefit was noted before the scheduled completion of the trial, hence; the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less